CLINICAL TRIAL: NCT00233064
Title: A Phase IV, Randomized, Double-Blind Study to Assess the Immune Reactivity of the Liquid and Lyophilized Formulations of Palivizumab (MEDI-493, Synagis) in Children at High Risk for the Development of Serious RSV Disease
Brief Title: Study to Assess the Immune Reactivity of the Liquid and Lyophilized Formulations of Palivizumab (MEDI-493, Synagis)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Genevieve Losonsky, M.D., MedImmune Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP116
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2008-10-28 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2010-01

CONDITIONS: Chronic Lung Disease
MeSH Terms: interventions — Palivizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Liquid Palivizumab
  Interventions: Biological: Liquid Palivizumab
- 2 (Active Comparator): Lyophilized Palivizumab
  Interventions: Biological: Lyophilized Palivizumab

INTERVENTIONS:
Biological: Lyophilized Palivizumab — Patients will receive 15 mg/kg of lyophilized palivizumab administered intramuscularly every 30 days for a total of 5 injections.
  Other Names: Synagis
  Arms: 2
Biological: Liquid Palivizumab — Patients will receive 15 mg/kg of liquid palivizumab administered intramuscularly every 30 days for a total of 5 injections.
  Other Names: Synagis
  Arms: 1

SUMMARY:
The purpose of this study is to measure the rate of anti-palivizumab antibodies (also referred to as immune reactivity or immunogenicity) in subjects receiving either the liquid or lyophilized formulation of palivizumab. This study will compare the number and percentage of subjects with anti-palivizumab antibodies receiving either the liquid or lyophilized formulation of palivizumab.

DETAILED DESCRIPTION:
The approved liquid formulation of palivizumab was developed to simplify preparation of the drug before injection. Both formulations of palivizumab have been shown to be bioequivalent in children 6 months of age or younger with a history of chronic lung disease. In previous studies of liquid palivizumab, immunogenicity was evaluated up to 2 months after dosing in adults, and 1 month after dosing in children. In this study, MI-CP116, immunogenicity will be evaluated between 4 and 6 months after the last dose of study drug, in order to provide data at a time point significantly distant from dosing when drug interference is minimal.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable child with chronic lung disease of prematurity who is ≤24 months of age at randomization OR child with premature birth (gestational age ≤35 weeks or less) and who is 6 months of age or younger at randomization
* Written informed consent obtained from the patient's parent(s) or legal guardian(s)
* The child must be able to complete the follow-up visit 4-6 months after the last dose of study drug

Exclusion Criteria:

* Hospitalization at the time of randomization (unless discharge is anticipated within 3 weeks)
* Be receiving mechanical ventilation at the time of study entry (including CPAP)
* Congenital heart disease (children with uncomplicated CHD [e.g., PDA, small septal defect] and children with complicated CHD who are currently anatomically and hemodynamically normal can be enrolled).
* Mother with HIV infection (unless the child has been proven to be not infected)
* Life expectancy <6 months
* Known allergy to Ig products
* Acute respiratory or other acute infection or illness
* Previous reaction to IGIV, blood products, or other foreign proteins
* Receipt of lyophilized palivizumab, RSV-IG IV, or other RSV-specific monoclonal antibody, or any other polyclonal antibody (for example, Hepatitis B IG, IVIG, VZIG) within 3 months prior to randomization
* Any previous receipt of MEDI-524
* Participation in other investigational drug product studies

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 417 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Genny Losonsky, MD, Study Director — MedImmune LLC
Locations (53):
- United States (53):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Clinical Research Consultants, Hoover, Alabama
  - The University of Alabama School of Medicine, Tuscaloosa, Alabama
  - All for Kids Pediatric Clinic, Little Rock, Arkansas
  - Family Medical Center, Foothill Ranch, California
  - Edinger Medical Group, Fountain Valley, California
  - Doctors Medical Group, West Covina, California
  - Convenience Care, West Covina, California
  - Norwich Pediatric Group, P.C., Norwich, Connecticut
  - The Allergy Center at Brookstone, Columbus, Georgia
  - Physicians to Children and Adolescents, Bardstown, Kentucky
  - Peak Medical Research LLC, Owensboro, Kentucky
  - Boston University Medical Center, Boston, Massachusetts
  - Pediatric Association of Fall River, Fall River, Massachusetts
  - Woburn Pediatric Associates, Woburn, Massachusetts
  - Michigan Institute of Medicine, Livonia, Michigan
  - Meridian Clinical Research, Omaha, Nebraska
  - St. Joseph's Childrens Hospital, Paterson, New Jersey
  - Maimonides Pediatric Pulmonology, Brooklyn, New York
  - North Carolina Children's & Adult's Clinical Research Foundation/Purcell Clinic, Laurinburg, North Carolina
  - Capitol Pediatric And Adolescent Center, Raleigh, North Carolina
  - North Carolina Children's and Adult's Clinical Research Foundation, Sylva, North Carolina
  - Medcenter One/Q&R Clinic, Bismarck, North Dakota
  - Dakota Clinic, Ltd. / Innvois Health, Fargo, North Dakota
  - Trinity Medical Group-Health Center Medical Arts, Minot, North Dakota
  - Dr. Shelly David Senders, M.D., Inc., Cleveland, Ohio
  - Northeast Cincinnati Pediatric Associates, Inc, Mason, Ohio
  - Santiago Reyes, M.D., Oklahoma City, Oklahoma
  - Tri-State Pediatrics, Beaver Falls, Pennsylvania
  - Greenville Medical Center, Greenville, Pennsylvania
  - CCP - Armstrong Pediatrics, Kittanning, Pennsylvania
  - Pediatric Alliance of Latrobe, Latrobe, Pennsylvania
  - Temple Univ. Children's Medical Center, Philadelphia, Pennsylvania
  - Pediatric Alliance, Southwestern, Pittsburgh, Pennsylvania
  - South Hills Pediatrics, Pittsburgh, Pennsylvania
  - Primary Physician's Research, Inc., Pittsburgh, Pennsylvania
  - Laurel Pediatrics, Uniontown, Pennsylvania
  - Brown Clinic P.L.L.P./Northridge Clinic, Watertown, South Dakota
  - Jackson Clinic, Jackson, Tennessee
  - Holston Medical Group; Pediatrics at Meadowview Lane, Kingsport, Tennessee
  - Holston Medical Group; Pediatrics at Stone Plaza, Kingsport, Tennessee
  - Sadler Clinic, Conroe, Texas
  - Pediatric Allergy/Immunology Associates, PA, Dallas, Texas
  - MedPro Research, Houston, Texas
  - Pediatric Associates, Houston, Texas
  - Quality Assurance Research Center, San Antonio, Texas
  - Wee Care Pediatrics, Layton, Utah
  - Bear Care Pediatrics, Ogden, Utah
  - Utah Valley Pediatrics, Provo, Utah
  - Families First Pediatrics, South Jordan, Utah
  - Advanced Pediatrics, Vienna, Virginia
  - WVU Department of Pediatrics, Charleston, West Virginia
  - Monroe Clinic, Monroe, Wisconsin

REFERENCES:
- [Background] Makari D, Jensen KM, Harris B, Jafri HS. Randomized, Double-Blind Study of the Safety of the Liquid Versus Lyophilized Formulation of Palivizumab in Premature Infants and Children with Chronic Lung Disease of Prematurity. Infect Dis Ther. 2014 Dec;3(2):339-47. doi: 10.1007/s40121-014-0033-y. Epub 2014 Aug 26. PMID 25156956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 417 subjects were randomized into the study at 51 sites in the United States between 20 October 2005 and 02 October 2007.
Pre-assignment Details: A total of 4 subjects at site #1022 who received all 5 doses of study drug (per drug accountability records) had no further information including case report form that could be obtained. These 4 subjects were excluded from all data analyses.
Groups:
- Liquid Palivizumab: Liquid Palivizumab, 15 mg/kg IM q30 days X 5
- Lyophilized Palivizumab: Lyophilized Palivizumab, 15 mg/kg IM q30 days X 5
Period: Overall Study
Arm/Group | Liquid Palivizumab | Lyophilized Palivizumab
Started | 211 | 202
Completed | 197 | 190
Not Completed | 14 | 12
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Death | 0 | 1
Not completed — Relocation | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Moved to Dom. Republic | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liquid Palivizumab | Lyophilized Palivizumab | Total
Number analyzed (Participants) | 211 | 202 | 413
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.56 (4.50) | 4.00 (4.16) | 4.29 (4.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 99 | 203
  Male | 107 | 103 | 210
Region of Enrollment [Number; unit: participants]
  United States | 211 | 202 | 413
Chronic Lung Disease at Prematurity [Number; unit: Participants]
  Yes | 35 | 26 | 61
  No | 176 | 176 | 352
Race/Ethnicity [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 24 | 49
  White | 151 | 149 | 300
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Hispanic | 22 | 14 | 36
  Other | 12 | 12 | 24
Gestational Age at Birth [Mean (Standard Deviation); unit: Weeks] | 32.4 (2.7) | 32.7 (2.5) | 32.5 (2.6)
Weight at Day 0 [Mean (Standard Deviation); unit: Kilogram] | 5.326 (2.274) | 5.079 (2.264) | 5.205 (2.270)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Immune Reactivity
Description: Presence of anti-palivizumab antibodies
Time Frame: Day 240-300 follow up
Population: Participants who received at least 2 doses of study drug and had at least 1 blood sample collected (at baseline or Study Day 240-300) were included in the analysis. This included 206 subjects in Arm 1 and 200 subjects in Arm 2. Of these subjects, 191 (Arm 1) and 188 (Arm 2) had adequate blood samples for analysis. This analysis was per protocol.
Measure: Number; unit: Participants
Arm/Group | Liquid Palivizumab | Lyophilized Palivizumab | Combined Liquid/Lyophilized Palivizumab
Number analyzed (Participants) | 191 | 188 | 379
Participants
  Number | 0 | 1 | 1
  Percentage | 0.0 | 0.5 | 0.3
Statistical Analysis 1: Comparison: Liquid Palivizumab; The subject number of 200 per treatment group was derived to demonstrate a percentage of immune reactivity in either the liquid or lyophilized formulations of palivizumab of <2-3% based on 95% confidence intervals [(0%; 0.00, 1.83), (0.5%; 0.01, 2.75), (1%; 0.12, 3.57)]; Test type: Superiority or Other; Overall percentage of immune reactivity = 0.0, 95% CI [0.0 to 1.9] — The number and percentage of subjects with immune reactivity at Study Day 240-300 were constructed using the Clopper-Pearson Method
Statistical Analysis 2: Comparison: Lyophilized Palivizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Overall percentage of immune reactivity = 0.5, 95% CI [0.0 to 2.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Combined Liquid/Lyophilized Palivizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Overall percentage of immune reactivity = 0.3, 95% CI [0.0 to 1.5] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time of the first study drug administration through Study Day 150. Adverse events were not collected in this study.
Arm/Group | Liquid Palivizumab | Lyophilized Palivizumab
Serious Adverse Events (participants affected / at risk) | 18/211 | 12/202
Other Adverse Events (participants affected / at risk) | 0/211 | 0/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liquid Palivizumab (N=211) | Lyophilized Palivizumab (N=202)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cleft Lip (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 6 (6) | 3 (3)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infectious Croup (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis Rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 2 (2) | 0 (0)
Occult Blood Positive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Craniosynostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Complex Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Convulsions (Nervous system disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Only serious adverse events were collected as part of the safety evaluation. One death (asphyxia) occurred in the Lyophilized Palivizumab group; this event was judged not related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.